CLINICAL TRIAL: NCT04985578
Title: Effects on Muscle Activity After Dry Needling in Myofascial Trigger Points of the Gastrocnemius Muscles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS-2018-11C
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Myofascial Trigger Point Pain
Keywords: dry needling; gastrocnemius; myofascial trigger point; Superficial Electromyography
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know if patients have received the dry needling technique or not.
  Participants in the sham group will told they will receive a normal dry needling protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling Group (Experimental): The experimental extremity will be assigned randomly and will receive a single treatment session of TrP dry needling as follows: the therapist will located the TrP that refers the most pain and will apply manual compression until the participant will reported pain. After that, dry needling technique will be performed on the TrP for 60 seconds.
  Interventions: Other: Dry needling
- Sham dry needling (Placebo Comparator): The experimental extremity will be assigned randomly and will receive a single treatment session of TrP sham dry needling as follows: the therapist will located the TrP that refers the most pain and will apply manual compression until the participant will reported pain. After that, sham dry needling technique will be performed on the TrP for 60 seconds with a needle without tip.
  Interventions: Other: Sham dry needling
- Control (No Intervention): No Treatment will be perfomed in this group

INTERVENTIONS:
Other: Dry needling — The therapist will located the TrP that refers the most pain and will apply manual compression until the participant will reported pain. After that, dry needling technique will be performed on the TrP for 60 seconds.
  Arms: Dry needling Group
Other: Sham dry needling — The therapist will located the TrP that refers the most pain and will apply manual compression until the participant will reported pain. After that, dry needling technique will be performed on the TrP for 60 seconds with a sham needle without tip.
  Arms: Sham dry needling

SUMMARY:
Trigger points (TrPs) are a common musculoskeletal cause of local and referred muscle pain, as well as local inflammation in the muscle and fascia. From a clinical and sensory viewpoint, TrPs may be classified as active or latent. The principal difference is the reproduction of symptoms experienced by an individual (active) with or without stimulation. Local and referred pain elicited from latent TrPs may be transient in duration upon stimulation, and latent TrPs may be present without spontaneous symptoms.

Both active and latent TrPs induce motor dysfunctions such as stiffness, restricted range of motion, and accelerated fatigability in the affected muscle. The interrater reliability of manual identification of latent TrPs in the calf muscles has been found to range from small to moderate. The clinical relevance of latent TrPs has increased in the last decade,4 and some studies have investigated the effects of treating them. Among all manual therapies targeted to latent TrPs, ischemic compression, or TrP pressure release, is the most commonly used. Although TrPs may affect any muscle, the gastrocnemius muscle may be the most susceptible in the lower extremity to developing them. It has been reported that 13% to 30% of the asymptomatic population has latent TrPs in these muscles, and their presence may affect sport practice.

The purpose of this study will be to evaluate changes in muscle activity in myofascial trigger points (TrPs) after a single treatment session of dry needling in the gastrocnemius muscle.

A randomized controlled clinical trial with blinded assessor will be conducted. 90 asymptomatic volunteers with MrPs gastrocnemius -muscle TrPs will bilaterally explored. After exploration the volunteer will be asigned to either Control (no treatment), experimental (60 seconds of dry needling on the TrP that refers more pain on the randomly assigned extremity) or sham group (60 seconds of dry needling on the TrP that refers more pain with a sham needle with no tip). To be part of the sham group patients should not have received any dry needling before.

Muscle activity is commonly recorded in research using surface electromyography (sEMG). sEMG has previously been used in similar studies because it is less invasive than intramuscular electromyography. Electromyography will be performed using the mDurance® surface electromyograph (mDurance Solutions SL; Granada, Spain) in order to capture muscle activity of the lateral and medial Gastrocnemius muscles (Electrodes will be placed as described by the mDurance application) during an unilateral countermovement Jump (in both extremities) and 20 meter Sprint. There will be a resting period of at least 2 minutes between exercises to prevent the results from being affected by fatigue.

ELIGIBILITY:
Inclusion Criteria:

* A TrP will be diagnosed using the following criteria: palpable taut band, presence of a painful spot in the taut band, and referred pain on palpation of the spot.

Exclusion Criteria:

* Participants were excluded if they reported any pain symptoms in the lower extremities in the previous year.
* They were also excluded if they presented previous surgical interventions, previous lower-extremity injury, any underlying medical disease, pregnancy, or muscle soreness after vigorous exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Muscle activity (microVolts) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  sEMG is a NON-invasive method that measures the electrical activity of the muscle generated by the passage of the nerve impulse, which causes depolarization of the muscle cell membrane during excitation. Once the muscle is contracted and receives electrical signals, the electrodes pick up these signals and record them on the device application.

SECONDARY OUTCOMES:
Jump Force (Newtons) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Jump Force will be measured using the Myjump app.
Jump Height (centimeters) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Jump Height will be measured using the Myjump app.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional Catalunya, Barcelona, Sant Cugat, Spain